CLINICAL TRIAL: NCT06219525
Title: Higher and Standard Doses of Enteral Zinc Supplementation in Very Preterm Infants: A Randomized Controlled Trial
Brief Title: Higher and Standard Doses of Enteral Zinc Supplementation in Very Preterm Infants
Acronym: ZnVeryPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Anucha Thatrimontrichai, Associated professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 66-451-1-1; 66-451-1-1 (Other Grant/Funding Number: Faculty of Medicine, Prince of Songkla University)
Record Dates: First submitted 2023-12-25; First posted 2024-01-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Very Preterm Infants; Zinc Deficiency
Keywords: Growth and Development; Mortality; Newborn; Premature Infant; Zinc
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The study design was approved by the ethics committee of our Center. Written informed consent was obtained from the parents of the infants enrolled in the study. Stratification was performed based on birthweight [BW] (401-999 or 1,000-1,499 or 1,500-1800 grams) and small for gestational age (yes or no). Participants were randomly allocated (1:1) to one of two treatments (higher or standard doses of zinc supplement). The allocation sequence was performed via computer generation, with permuted block and kept as consecutive numbers by statistician. Allocation concealment was ensured by using identical, opaque, and sealed envelopes.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The two doses of zinc preparations were provided in identical bottles without indication of group identity or content by a neonatal registered pharmacist (assigned participants to interventions, only unblinded investigator) in the study center. A dedicated nurse (enrolled participants, obtained informed consent, monitored intervention, and recorded data), registered nurses and attending neonatologists (did routine neonatal care), statistician (generated the allocation sequence), and dedicated clinical psychologist were blinded the allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher dose of enteral zinc (Active Comparator): higher dose of zinc sulfate 10 mg/day; each 1 mL contains 10 mg of elemental zinc (osmolality 450 Osm/kg H2O).
  Interventions: Dietary Supplement: Higher dose of enteral zinc
- Standard dose of enteral zinc (Placebo Comparator): standard dose of zinc sulfate 1 mg/day; each 1 mL contains 1 mg of elemental zinc (osmolality 45 Osm/kg H2O).
  Interventions: Dietary Supplement: Standard dose of enteral zinc

INTERVENTIONS:
Dietary Supplement: Higher dose of enteral zinc — Higher dose of zinc sulfate 10 mg/day; each 1 mL contains 10 mg of elemental zinc (osmolality 450 Osm/kg H2O). After randomization, nurses blinded to the study aims administered the assigned preparation 1 mL via tuberculin syringe, once daily, 1 hour after feeding. Zinc sulphate oral solution was prepared by the pharmaceutical compounding unit in the hospital. The supplement was given again to subjects who vomited within 15 minutes after the administration. All episodes of vomiting were reported on the record form. Vomiting episodes within 15 minutes were recorded. The supplement assigned was at discharge or at 44 weeks of postmenstrual age whichever came first. Both groups received multivitamin (MTV) products and iron supplement as routine preterm care.
  Arms: Higher dose of enteral zinc
Dietary Supplement: Standard dose of enteral zinc — Standard dose of zinc sulfate 1 mg/day; each 1 mL contains 1 mg of elemental zinc (osmolality 45 Osm/kg H2O). After randomization, nurses blinded to the study aims administered the assigned preparation 1 mL via tuberculin syringe, once daily, 1 hour after feeding. Zinc sulphate oral solution was prepared by the pharmaceutical compounding unit in the hospital. The supplement was given again to subjects who vomited within 15 minutes after the administration. All episodes of vomiting were reported on the record form. Vomiting episodes within 15 minutes were recorded. The supplement assigned was discontinued at discharge or at 44 weeks of postmenstrual age whichever came first. Both groups received multivitamin (MTV) products and iron supplement as routine preterm care.
  Arms: Standard dose of enteral zinc

SUMMARY:
The goal of this randomized clinical trial is to compare the effect of higher (10 mg per day) versus standard (1 mg per day) doses of zinc supplementation The main questions it aims to answer are:

* Growth velocities and delta z-scores during the date of start intervention until the end of the time interval (at least 2 weeks of intervention on date of 44 weeks of postmenstrual age or discharge whichever came first) in very preterm infants with a birthweight less than1800 grams.
* Growth and neurodevelopment at 24 months postnatal age

DETAILED DESCRIPTION:
After informed consent, the neonates enrolled were randomly allocated to two study groups: group A (higher dose of zinc sulfate 10 mg/day; each 1 mL contains 10 mg of elemental zinc; Pharmacy Division, Songklanagarind Hospital), and group B (standard dose of zinc sulfate 1 mg/day; each 1 mL contains 1 mg of elemental zinc; Pharmacy Division, Songklanagarind Hospital).

The zinc solution was available as a white powder in white opaque plastic container. When normal sterile water was added up to the indicator mark, it provided 60 mL of solution containing 10 mg/mL (osmolality 450 Osm/kg H2O) and 1 mg/mL (osmolality 45 Osm/kg H2O) of elemental zinc with similar color, taste and packing. The two doses of zinc preparations were provided in identical bottles and was labeled only zinc solution, hospital number and name-surname, without indication of group identity (A or B) or concentration by a neonatal registered pharmacist in the study center (only unblinded investigator who recorded the group allocation according to the randomization list in consecutive participant). This information was not available to the investigators during the data had been obtained, entered in the database, and analyzed by a blinded statistician.

After randomization, nurses blinded to the study aims administered the assigned preparation 1 mL via tuberculin syringe, once daily, 1 h after feeding. Zinc sulphate oral solution was prepared by the pharmaceutical compounding unit in the hospital. Each subject received a 60-mL bottle solution individually and continued the medication until finished, either at a concentration of 1 or 10 mg/mL, depending on the study group. The supplement was given again to subjects who vomited within 15 min after the administration. All episodes of vomiting were reported on the record form. Vomiting episodes within 15 min were recorded. The supplement assigned was discontinued at discharge or at 44 weeks' postmenstrual age whichever came first. Both groups received multivitamin products (1 mL/day) and iron supplement (2-3 mg/kg/day) as routine preterm care.

ELIGIBILITY:
Inclusion Criteria:

* Very preterm neonates (gestational age [GA]: 24 0/7-32 6/7 weeks and BW: 401-1800 grams) were consecutively admitted in the NICU and NMCU
* Body weight at enrollment less than 800 grams
* Stable neonates and full enteral feeding (150 mL/kg/day) at least for a few days

Exclusion Criteria:

* Outborn neonate who was admitted in study center after 7 days of life
* Congenital infections
* Malformations, syndromes, or genetic defects
* Evidence of culture proven sepsis or necrotizing enterocolitis or death diagnosed before enrollment
* Gastrointestinal (GI) surgery or high GI fluid output (usually ileostomy losses)
* Unstable neonate during weighing including on intercostal drainage tube or drainage
* Neonates need diuretics more than 7 days
* Severe birth asphyxia (5-minute Apgar score less than 4)
* Parents' decision not to participate the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight velocity during the date of start intervention until the end of the time interval (at least 2 weeks of intervention on date of 44 weeks of postmenstrual age or discharge whichever came first) | during the date of start intervention until the end of the time interval (at least 2 weeks of intervention on date of 44 weeks of postmenstrual age or discharge whichever came first)
  Weight velocity was calculated during the beginning of study (time1 [T1], Weight1 [W1]) until the end of the time interval (time2 [T2], Weight [W2]). Weight gain (grams per kilogram per day) was calculated during the period using the 2-point average method [1000*(W2-W1)]/[(W2+W1)/2)*(T2-T1)].
  Weight delta z-scores of were calculated weight z-scores at T2 minus weight z-scores at T1 from the Fenton's Growth Chart
Length velocity during the date of start intervention until the end of the time interval (at least 2 weeks of intervention on date of 44 weeks of postmenstrual age or discharge whichever came first) | during the date of start intervention until the end of the time interval (at least 2 weeks of intervention on date of 44 weeks of postmenstrual age or discharge whichever came first)
  Length velocity was calculated during the beginning of study (time1 [T1], Length1 [L1]) until the end of the time interval (time2 [T2], Length [L2]). Length velocities (centimeters per kilogram per day) was calculated during the period using the 2-point average method [1000*(L2-L1)]/[(L2+L1)/2)*(T2-T1)] Length delta z-scores were calculated length z-scores at T2 minus length z-scores at T1 from the Fenton's Growth Chart
Head circumference (HC) velocity during the date of start intervention until the end of the time interval (at least 2 weeks of intervention on date of 44 weeks of postmenstrual age or discharge whichever came first) | during the date of start intervention until the end of the time interval (at least 2 weeks of intervention on date of 44 weeks of postmenstrual age or discharge whichever came first)
  HC velocity was calculated during the beginning of study (time1 [T1], HC1) until the end of the time interval (time2 [T2], HC2). HC velocities (centimeters per kilogram per day) was calculated during the period using the 2-point average method [1000*(HC2-HC1)]/[(HC2+HC1)/2)*(T2-T1)] HC delta z-scores were calculated HC z-scores at T2 minus HC z-scores at T1 from the Fenton's Growth Chart

SECONDARY OUTCOMES:
Growth at 24 months postnatal age (PNA) | At 24 months PNA (20-24 months corrected age)
  Growth [at 24 months PNA, 20-24 months corrected age]) was assessed by corrected age
Neurodevelopment at 24 months postnatal age (PNA) | At 24 months PNA (20-24 months corrected age)
  Neurodevelopmental outcomes (Bayley-III tests, were evaluated by only dedicated clinical psychologists at 24 months PNA [20-24 months corrected age]) were assessed by corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Anucha Thatrimontrichai, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Sahin S, Sari FN, Bidev D, Bozkurt O, Dizdar EA, Oguz SS. Zinc Supplementation in Very Low Birth Weight Infants: A Randomized Controlled Trial. Am J Perinatol. 2024 May;41(S 01):e3107-e3114. doi: 10.1055/s-0043-1776762. Epub 2023 Nov 8. PMID 37939725
- [Background] Ram Kumar TV, Ramji S. Effect of zinc supplementation on growth in very low birth weight infants. J Trop Pediatr. 2012 Feb;58(1):50-4. doi: 10.1093/tropej/fmr036. Epub 2011 May 5. PMID 21546443
- [Background] Terrin G, Berni Canani R, Passariello A, Messina F, Conti MG, Caoci S, Smaldore A, Bertino E, De Curtis M. Zinc supplementation reduces morbidity and mortality in very-low-birth-weight preterm neonates: a hospital-based randomized, placebo-controlled trial in an industrialized country. Am J Clin Nutr. 2013 Dec;98(6):1468-74. doi: 10.3945/ajcn.112.054478. Epub 2013 Sep 11. PMID 24025633